CLINICAL TRIAL: NCT00251797
Title: A Phase I Trial Using Combination Irinotecan and Thalidomide for Recurrent CNS Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Dennie Jones, MD, University of New Mexico CRTC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2799C
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2008-10

CONDITIONS: Brain and Nervous System; Cancer
Keywords: Phase I; Brain cancer; Recurrent CNS tumors
MeSH Terms: conditions — Neurologic Manifestations; Neoplasms; Brain Neoplasms; Central Nervous System Neoplasms | interventions — Irinotecan; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Irinotecan — Irinotecan: 300 to 350 mg/m2 mixing with 250 cc. Dextrose injection. IV infusion over 90 minutes D1 and repeat every 21 days
  Other Names: Camptosar
Drug: Thalidomide — Thalidomide 50 mg capsule starting from 4 tablets per day Oral D 3 to D 19 of each cycle
  Other Names: Thalomid

SUMMARY:
The study will try to answer these questions:

1. What is the highest dose of thalidomide brain cancer patients can receive safely in combination with irinotecan?
2. How well does this combination work to shrink brain tumors, and how long do responses to treatment last?
3. What side effects does the combination of drugs cause?
4. How does treatment affect patients' quality of life (how they feel and what activities they are able to do)?

DETAILED DESCRIPTION:
This is a Phase I study, which means these trials are generally comparatively small and are used to determine toxicity and maximum dose. Currently, there are no "standard" treatments for Recurrent CNS Tumors. In this study, approximately 14 patients with Recurrent CNS Tumors will receive treatment with irinotecan, an intravenous drug, and thalidomide, a drug taken by mouth. Both have been approved by the Federal Food and Drug Administration as treatments for cancer, but they have not been tested together for brain cancer.

The study will try to answer these questions:

1. What is the highest dose of thalidomide brain cancer patients can receive safely in combination with irinotecan?
2. How well does this combination work to shrink brain tumors, and how long do responses to treatment last?
3. What side effects does the combination of drugs cause?
4. How does treatment affect patients' quality of life (how they feel and what activities they are able to do)?

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven high grade astrocytomas, glioblastoma multiforme, anaplastic astrocytoma, anaplastic oligodendroglioma, mixed oligodendroglioma.
* Subjects are allowed to have definitive surgery and/or radiation treatment to their tumors.
* Subjects are allowed to have previous chemotherapy for their tumors.
* Subjects who previous diagnosed to have a low grade lesion need a second biopsy to show transformation into a high grade histology.
* Subjects need to have radiographic or biopsy proven recurrent disease.
* ECORT performance status 2 or lower. See appendix I.
* Baseline laboratory values within 30 days of study entry: hemoglobin 10 gm/dl; absolute neutrophil count 1,500 cells/ml; platelet counts 100,000 cells/ml; SGOT/AST, SGPT/ALT, alkaline phosphatase, LDH 3high normal limit; total bilirubin 2.0 mg/dl.
* Ability to provide written informed consent.
* Age > 18 years.
* Female patients of childbearing potential must have a documented negative serum pregnancy test within 14 days of study entry.
* All subjects must agree to use an effective method of contraception for the duration of treatment if engaged in sexual activity where conception is possible, as specified in the STEP program for thalidomide.

Exclusion Criteria:

* Therapy with any investigational drug (other than drugs available on treatment IND and used for FDA-sanctioned indications) and/or any chemotherapy regimen within 28 days of study entry.
* Prior therapy with either irinotecan or thalidomide.
* Oxygen saturation 90% on room air.
* Cardiac insufficiency at New York Heart Association status 2 or greater.
* Other active malignancies except basal or squamous cell carcinoma of the skin or in situ cervical and breast lesions.
* History of neuropsychiatric disorder or altered mental status which prevent informed consent or compliance with protocol requirement.
* Known hypersensitivity or allergic reaction to study drug.
* Women at any stage of pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2000-03; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Tolerable dosage of thalidomide in combination with irinotecan | Unacceptable toxicities

SECONDARY OUTCOMES:
Tumor response. For this study, the definition of response will include complete response, partial response and stable disease. Duration of tumor response. uality of life while on treatment | unacceptable toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Dennie Jones, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States